CLINICAL TRIAL: NCT06840171
Title: The Effect of Mandala Coloring on Depression, Anxiety and Quality of Life of Inpatients in a Psychiatric Clinic
Acronym: Mandala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: reyhan eskiyurt (Other)
Responsible Party: Sponsor-Investigator, reyhan eskiyurt, Director, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YBU-378
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (mandala coloring) (Experimental): Mandala group will participate in 8 sessions of mandala application. Mandala Coloring Application will be applied to the Intervention group 2-3 times a week for 3 weeks. Mandala application will be done by the researcher and feedback about the mandala will be received from the patients at the end of each session. Data collection forms will be applied before the mandala painting application starts and after the mandala painting application ends (after the 8th session).
  Interventions: Other: Mandala coloring
- Control (No Intervention): No intervention will be applied to the patients in the control group during the follow-up period, only data collection forms will be applied.

INTERVENTIONS:
Other: Mandala coloring — Mandala group will participate in 8 sessions of mandala application. Mandala Coloring Application will be applied to the Intervention group 2-3 times a week for 3 weeks. Mandala application will be done by the researcher and feedback about the mandala will be received from the patients at the end of each session. Data collection forms will be applied before the mandala painting application starts and after the mandala painting application ends (after the 8th session).
  Arms: Experimental (mandala coloring)

SUMMARY:
The aim of this study is to examine the effects of mandala coloring activity applied to individuals hospitalized in a psychiatric clinic with a diagnosis of anxiety and depression disorder on quality of life, psychological resilience and depression, anxiety and stress levels.

DETAILED DESCRIPTION:
Introduction: It is stated that healthcare professional-patient interaction and patient activity improve clinical outcomes for patients with mental illness. When compared to psychosocial interventions, the most commonly used method in 49% of clinics was found to be artistic practices. It is stated that mandala painting has a calming and healing effect on the individual, facilitating psychological integration and personal meaning in life.

Objective: The aim of this study is to examine the effects of mandala coloring activity applied to individuals hospitalized in a psychiatric clinic with a diagnosis of anxiety and depression disorder on quality of life, psychological resilience and depression, anxiety and stress levels.

Method: The research will be conducted using a randomized controlled experimental research design. The research sample will consist of 50 patients in a university hospital psychiatry clinic. Research data will be collected using the Introductory Information Form, Depression-Anxiety-Stress Scale Short Form, Quality of Life Scale (SF-12), and Brief Resilience Scale. Patients diagnosed with anxiety and depression will undergo 8 sessions of mandala application. Data will be collected in two time periods before starting the mandala application and at the end of the 8-session application.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Being 18 years of age or older
* Diagnosed with anxiety and depression disorder

Exclusion Criteria:

* Those who gave incomplete answers to the scales used in the study
* Those with serious psychiatric symptoms (e.g. harming themselves or others, sedation)
* Those who did not participate in the mandala coloring session
* Those who did not agree to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-02-22 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Depression-Anxiety-Stress Scale | 3 week
  The scale, developed to determine the depression, anxiety and stress levels of individuals, consists of 21 items and 3 subscales. Depression-Anxiety-Stress Scale is a 4-point Likert-type measurement tool (0-not suitable for me and 3-completely suitable for me). The Turkish validity and reliability study of Depression-Anxiety-Stress Scale was conducted. High scores on the scale reveal which of the depression, anxiety and stress sub-dimensions the individual is experiencing problems with.
Quality of Life Scale | 3 week
  Quality of life scale (The SF-12) has two summary scales: physical component and mental component. The physical component summary scale consists of physical function, physical role, body pain and general health subscales, and the mental component summary consists of vitality, social function, emotional role and mental health subscales. The score of each subscale varies between 0-100 and the score is directly proportional to the quality of life. The Turkish validity and reliability study of the scale was conducted. Minimum and maximum scores can range from 0-100 from the scale. High scores indicate high quality of life.
Brief Psychological Resilience Scale | 3 week
  Brief Psychological Resilience Scale is a 5-point Likert-type, 6-item, self-report measurement tool. After the reverse-coded items in the scale are translated, high scores indicate high psychological resilience. The Turkish validity and reliability study of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Eskiyurt, Study Director — Yıldırım Beyazıt U
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)